CLINICAL TRIAL: NCT04801563
Title: Allogeneic Transplantation in Patients With Myelodysplastic Syndrome Based on Risk According to Revised-International Prognostic Scoring System (R-IPSS)
Brief Title: Allogeneic HSCT in MDS Patients Based on Risk According to R-IPSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Andrea Velardi, FULL PROFESSOR, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03/19
Record Dates: First submitted 2021-02-28; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: MDS and Allogeneic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SINGLE ARM (Other)
  Interventions: Other: MDS and AlloHSCT

INTERVENTIONS:
Other: MDS and AlloHSCT — Allogeneic stem cell transplantation, based on TMLI and followed by infusion of donor regulatory T cells and conventional T cells and purified donor CD34+ hematopoietic stem cells

SUMMARY:
An "intention-to-treat" study to evaluate the impact of allogeneic HSCT with Total Marrow and Lymphoid irradiation (TMLI), followed by Treg/Tcon adoptive immunotherapy, on overall survival in patients affected by Myelodysplastic Syndrome (MDS), according to IPSS-R.

DETAILED DESCRIPTION:
MDS patients with Intermediate, High, or Very-High R-IPSS risk will be enrolled. Allogeneic stem cell transplantation with regulatory and conventional T cell adoptive immunotherapy will be proposed to eligible High and Very-High risk MDS patients. Intermediate risk MDS patients will be assessed for risk modification every six months and moved to transplant in case of increased risk. Intermediate risk MDS patients will be also evaluated for the presence of molecular alterations (TP53, ASXL1, RUNX1). Overall survival of the entire cohort will be assessed as primary endpoint. Incidence of Treatment Related Mortality, acute Graft versus Host Disease, chronic Graft versus Host Disease, Relapse will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Myelodysplastic Syndrome with IPSS-R INT, HIGH or VERY HIGH;
* Age <71 years;
* Signature of the informed consent.

Exclusion Criteria:

* Patients affected by Myelodysplastic Syndrome with IPSS-R VERY LOW or LOW;
* Patients affected by Myelodysplastic Syndrome/Myeloproliferative Neoplasm;
* Age >70 years;
* No signature of the informed consent

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
overall survival | 4 years
  We will evaluate overall survival in patients with intermediate/High/very-High risk MDS

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Velardi, MD, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Perugia, PG, Italy

REFERENCES:
- [Result] Di Ianni M, Falzetti F, Carotti A, Terenzi A, Castellino F, Bonifacio E, Del Papa B, Zei T, Ostini RI, Cecchini D, Aloisi T, Perruccio K, Ruggeri L, Balucani C, Pierini A, Sportoletti P, Aristei C, Falini B, Reisner Y, Velardi A, Aversa F, Martelli MF. Tregs prevent GVHD and promote immune reconstitution in HLA-haploidentical transplantation. Blood. 2011 Apr 7;117(14):3921-8. doi: 10.1182/blood-2010-10-311894. Epub 2011 Feb 3. PMID 21292771
- [Result] Martelli MF, Di Ianni M, Ruggeri L, Falzetti F, Carotti A, Terenzi A, Pierini A, Massei MS, Amico L, Urbani E, Del Papa B, Zei T, Iacucci Ostini R, Cecchini D, Tognellini R, Reisner Y, Aversa F, Falini B, Velardi A. HLA-haploidentical transplantation with regulatory and conventional T-cell adoptive immunotherapy prevents acute leukemia relapse. Blood. 2014 Jul 24;124(4):638-44. doi: 10.1182/blood-2014-03-564401. Epub 2014 Jun 12. PMID 24923299